CLINICAL TRIAL: NCT01995396
Title: Hartmanns Procedure or Abdominoperineal Excision With Intersphincteric Dissection in Rectal Cancer: a Randomized Study
Acronym: HAPIrect
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision after interims analysis
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Kenneth Smedh, Professor, Region Västmanland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTV-398121
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Rectal Cancer; Sphincter Ani Incontinence; Other Diagnoses, Comorbidities, and Complications
Keywords: rectal cancer,; fecal incontinence,; severe co-morbidity,; Hartmann´s procedure,; abdominoperineal excision with intersphincteric dissection,; postoperative complications,; pelvic abscess,; perineal infections
MeSH Terms: conditions — Rectal Neoplasms; Fecal Incontinence; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- APE with intersphincteric dissection (Active Comparator): Abdominoperineal excision with intersphincteric dissection and a stoma is performed in patients with rectal cancer and fecal incontinence and/or severe co-morbidity
  Interventions: Procedure: Hartmann´s procedure
- Hartmann´s procedure (Active Comparator): Hartmann´s operation and stoma is performed in patients with rectal cancer and fecal incontinence and/or severe co-morbidity
  Interventions: Procedure: APE with intersphincteric dissection

INTERVENTIONS:
Procedure: APE with intersphincteric dissection — Abdominal operation where the rectum is resected down to the levator and then the anus is resected by an intersphincteric dissection and order to leave the outer sfincter and levator in place to avoid a large wound and a high rate of infectious complications.
  Arms: Hartmann´s procedure
Procedure: Hartmann´s procedure — Abdominal operation where the rectum is resected and stapled off distally and a stoma is created
  Arms: APE with intersphincteric dissection

SUMMARY:
In patients with rectal cancer, an anterior resection with a colo-rectal or colo-anal anastomoses is the gold standard. However, in patients with a weak sphincter and fecal incontinence or in patients with severe co-morbidity and reduced general condition, this operation is not suitable.

In these situations there are two other radical surgical options, Hartmanns procedure and the Abdominoperineal excision that can be performed with intersphincteric dissection to minimise perineal complications.There are no data on which of these procedures that are best suited for these patients with fecal incontinence or severe co-morbidity( at risk for life-threatening anastomotic leak). In this randomized study we intend to compare postoperative complications within 30 days after these two procedures and also late complications and quality of life after one year postoperatively.

DETAILED DESCRIPTION:
In patients with rectal cancer, an abdominal operation with anterior resection with total mesorectal excision is the gold standard. Colon is anastomosed to the ano-rectum.The potential risks are bad bowel function with fecal incontinence or a lifethreatening anastomotic dehiscence, especially in patients with severe co-morbidity or reduced general condition.Tumours in the low rectum are usually treated with an abdominoperineal resection where the whole anus is radically excised and a permanent colostomy is created.

For patients with incontinence and/or severe comorbidity, Hartmann´s procedure has often been performed. The rectum is resected, the lower part is transected with a stapler and a colostomy is created. During recent years there has been reports on high rates of pelvic abscesses after Hartmann´s. An alternative has been proposed, namely the abdominoperineal excision (APE) with intersphincteric dissection leaving the outer sphincter and levator muscles in place, thus creating a much lesser perineal wound that also tend to heal better when the ano-pelvic muscles are left in place.

There have been some small retrospective studies comparing postoperative complications after Hartmann´s with anterior resections or the classic abdominoperineal excision. These studies are heterogenous and not balanced and no conclusions can be drawn. There are no data on APE with intersphincteric dissection in rectal cancer patients.

There is a need to clarify what procedure is most suited for patients with rectal cancer and fecal incontinence and / or severe comorbidity.

For this patient group we intend to randomize between Hartmann´s procedure and APE with intersphincteric dissection.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer 5cm or more from the anal verge
* Both procedures should be possible to perform
* Patients should have co-morbidities and/or have weak anal sphincter where an anterior resection is not suitable
* Metastases are no contraindication but the procedure should be assessed as locally radical.
* Patients should be assesed to cope with a major abdominal procedure(ASA I-III)

Exclusion Criteria:

* rectal cancer below 5cm from the anal verge where a Hartmann is considered not to be locally radical.
* patients where an anterior resection is suitable
* ASA IV or worse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2014-02; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Rates ot postoperative surgical complications within 30 days. | 30 days
  Perineal and abdominal wound infection, pelvic abscess urinary catheter at discharge etc

SECONDARY OUTCOMES:
Peroperative data | day of surgery
  time of surgery, bleeding in ml, peroperative complications, type of staplers used
The rate of intraoperative perforations | day of surgery
  record perforation of rectum or tumour during surgery
Resection margins | 2-4 weeks after surgery
  Histopathological report
Rate of local recurrence | 3 and 5 years postoperatively
  Record local recurrence during follow-up. CT-scan after 1 and 3 years
Survival after 3 and 5 years follow-up | 3 and 5 years postoperativelly
  overall survival
Postoperative actions | within 30 days
  reoperation, interventions(percutaneous drains etc) hospital stay, rehospitalisation
Other postop complications | 30 days
  other infectious, cardio-pulmonary and thromb-embolic complications.

OTHER OUTCOMES:
quality of life between the two methods | Preoperative and one year after surgery
  QoL protocol according to the QoLiRECT-study (Quality of life rectal cancer study) a study running from Gothenburg, Sweden
Late complications after surgery | One year postoperativelly
  Perineal pain, secretion from the ano-rectal stump

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Smedh, PhD, Principal Investigator — Region Vastmanland
Locations (1):
- Västmanlands Hospital Västerås, Västerås, Sweden

REFERENCES:
- [Derived] Nikberg M, Akerlund V, Swartling T, Buchwald P, Smedh K; HAPIrect Collaborative Study Group. Postoperative complications in Hartmann's procedure versus intersphincteric abdominoperineal excision in rectal cancer: randomized clinical trial (HAPIrect). BJS Open. 2025 Sep 8;9(5):zraf093. doi: 10.1093/bjsopen/zraf093. PMID 41026509
- [Derived] Smedh K, Sverrisson I, Chabok A, Nikberg M; HAPIrect Collaborative Study Group. Hartmann's procedure vs abdominoperineal resection with intersphincteric dissection in patients with rectal cancer: a randomized multicentre trial (HAPIrect). BMC Surg. 2016 Jul 11;16(1):43. doi: 10.1186/s12893-016-0161-2. PMID 27401339